CLINICAL TRIAL: NCT03087357
Title: The VALUE Study - Women & Infants as the Coordinating Center
Brief Title: VAlidation of a Lower Cost aneUploidy scrEen
Acronym: VALUE
Status: Completed | Type: Observational
Sponsor: Women and Infants Hospital of Rhode Island (Other)
Collaborators: PerkinElmer, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 940244
Record Dates: First submitted 2017-03-01; First posted 2017-03-22 (Actual); Last update posted 2022-09-22 (Actual); Status verified 2022-09

CONDITIONS: Down Syndrome; Trisomy 18; Trisomy 13
MeSH Terms: conditions — Down Syndrome; Trisomy 18 Syndrome; Trisomy 13 Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Residual plasma samples, only with permission of enrolled women
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Low Risk: The Low Risk group will consist of 2,400 pregnancies with no high risk findings (e.g., abnormal ultrasound, positive serum screen) who are undergoing initial clinical cfDNA screening. To simulate a general pregnancy population, approximately 20% of these women will be age 35 and older. An estimated 2% (48) of these LR women will have a failed/no call cfDNA test. Consenting women will provide samples for SmartNIPT testing.
  Interventions: Other: SmartNIPT
- High Risk: The High Risk group will consist of 250 women with a positive cfDNA screen reported by a Clinical Laboratory Improvement Amendments (CLIA)-approved commercial laboratory, and who present for consideration of a confirmatory diagnostic test, (i.e., CVS or amniocentesis). Consenting women will provide samples for SmartNIPT testing.
  Interventions: Other: SmartNIPT

INTERVENTIONS:
Other: SmartNIPT — A novel, non-next generation sequencing (NGS) test that is designed to perform as well as conventional NGS screening while being simpler and less expensive.

SUMMARY:
This study will document the detection rate and false positive rate as well as failure rate of a new prenatal screening approach ('Smart NIPT') as described at www.vanadisdx.com and implemented in an academic laboratory with limited molecular testing experience. Testing will be performed on samples from a general risk pregnancy population, with additional high-risk cases added to improve confidence in the detection rate. Additional characteristics of this non-NGS test such as turn-around time, costs (equipment, training, per test), results reporting, fetal sex, fetal fraction, and quality measures will also be examined.

DETAILED DESCRIPTION:
Women & Infants Hospital of Rhode Island (WIH) will serve as the Study Center and the Laboratory Site. Enrollment Sites will secure local IRB approval, identify, consent and enroll pregnant women, ship plasma samples to WIH and collect outcome information. Eligible patients will be from one of two groups:

* The 'high risk' (HR) group - 250 women considering diagnostic testing, nearly all following a positive cell free (cf)DNA screening test. At least one case of Down syndrome should be detected for every three women enrolled, in addition to an occasional case of T18 or T13.
* The 'low risk' (LR) group - 2,400 women having conventional cfDNA screening as their primary screening test (i.e., no serum/ultrasound testing), representing the general pregnancy population. Their group risk of Down syndrome should be about 1:500. This group should have no more than 20% women age 35 and older. (Women whose conventional cfDNA screen is positive would then be eligible for a second enrollment in the 'high risk' group).

Both groups of women will be asked to provide three full 10mL Streck tubes of blood (two tubes minimum), agree to release limited clinical information, provide signed consent (including for FDA personnel to review records) and consent to have Enrollment Site staff review and report needed information from newborn/infant examination records, if requested. Identifiable patient information will be held at Enrollment Sites and not released to the Laboratory or Study Center. Sample and outcome information will be identified only by a unique study code. Individual cfDNA test results will not be returned to the Enrollment Sites, providers, or enrolled women. Enrollment Sites will receive a summary of results once the study ends.

Enrollment Sites are likely to enroll either HR or LR women, although a few sites may be able to enroll both. Both settings will have genetic counselors, physicians, research assistants or other medical staff available to identify, inform, consent and enroll women, as well as to collect and ship samples and obtain pregnancy outcome information. Staff designated as participating in the VALUE Study will be qualified to inform eligible women of the study's benefits and harms, and collect/document informed consent (which will remain at that site). The Study Center may request confirmation of consent, should it become necessary. Outcomes for HR women choosing diagnostic testing will be the results of the karyotype; those declining diagnostic testing will have newborn/infant information collected( often a newborn karyotype). In the LR population, a negative cfDNA test result will be accepted as ruling out a common autosomal trisomy, as the residual risk would be very low (<1:20,000 to < 1:50,000). For LR women with a positive cfDNA test, results of diagnostic testing would be requested. If diagnostic test results are unavailable, a review of the newborn examination/karyotype will be required for confirmation. Any conflicting results between the clinical tests and the VALUE Study results(false positive / false negative) would also require resolution that may involve review of newborn/infant records.

The VALUE Study intends to enroll approximately 2,400 LR women through as many as 8 LR Enrollment Sites associated with general risk obstetrical care practices. The 2,400 target is set to: 1) provide a reasonably confident estimate of an expected low false positive rate (e.g., 0.2%) and 2) provide sufficient numbers to exercise the testing platform over a 12 month time period. The target of 2,400 is large enough to meet both objectives and is slightly more than the largest number of euploid samples tested in any of the original NGS HR cfDNA validation studies (2011-2012). The number of trisomies detected in this LR group should be fewer than 10.An estimated 2% (48) of these LR women will have a failed/no call cfDNA test..

Sample handling:

Plasma samples could be tested fresh or stored and tested once the assay system has been validated. Outcome information will not be collected from Enrollment Sites until samples have been tested, ensuring blinding of laboratory to outcomes.

Timeframe:

Identification of Enrollment Sites and securing Investigational Review Board (IRB) approval will take three months. Efforts related to set-up and qualification of the testing laboratory is expected to take four to six months as will study-specific software development. Active enrollment is scheduled for 12 months. The intent is to run the majority of samples fresh, allowing for long-term assay variability to be studied. Follow-up will be completed, for the most part, within two months of the final testing (except for the small proportion of women who tested positive but did not have diagnostic testing). These will have outcomes confirmed at the time of delivery.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years old
* 10-20 weeks gestation

  * Low Risk group
* no known aneuploidy risk
* scheduled for cfDNA screen as primary aneuploidy screen

  * High Risk group
* positive cfDNA screen
* scheduled to discuss CVS/amniocentesis as confirmatory test

Exclusion Criteria:

* Triplet or higher order pregnancy

  * Low Risk group
* positive nuchal translucency (NT) or abnormal ultrasound
* previous pregnancy with aneuploidy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 1. Pregnant women who either have no known risk factors for fetal aneuploidy (Low Risk group) and who present for cfDNA screening as their primary screen at a qualified Enrollment Site.
  2. Pregnant women who have had a positive cfDNA screen and who present for discussion of confirmatory diagnostic testing (High Risk group) at a qualified Enrollment Site.
Sampling Method: Non-Probability Sample
Enrollment: 2443 (Actual)
Dates: Start 2017-10-10 (Actual); Primary Completion 2019-11-19 (Actual); Study Completion 2020-10-01 (Actual)

PRIMARY OUTCOMES:
Down syndrome detection rate | Karyotype at chorionic villous sampling (CVS)/amniocentesis within 48 hours of enrollment OR at examination of products of conception if fetal loss up to 30 weeks post enrollment OR at newborn examination 24-48 hours after birth
  The cfDNA test detection rate for Down syndrome will utilize both the general population (low risk) enrollment (2,400 pregnancies) as well as the high risk enrollment (250 pregnancies, all confirmed trisomy 21/18/13) and be defined as TP/(TP+FN). All low risk women with a cfDNA test positive for trisomy 21 will have comprehensive diagnostic follow-up as will all high risk women, assuring that all affected pregnancies in these two groups will have karyotype confirmation. The true positive (TP) SmartNIPT cfDNA test results will be positive and agree with the abnormal karyotype finding. The false negative (FN) SmartNIPT cfDNA test results will be negative for the abnormal karyotype finding.
Down syndrome false positive rate | Karyotype at chorionic villous sampling (CVS)/amniocentesis within 48 hours of enrollment OR at examination of products of conception if fetal loss up to 30 weeks post enrollment. OR negative newborn examination 24-48 hours after birth
  The false positive rate for Down syndrome will be computed using data from the general population (low risk) enrollment only (2,400 pregnancies) and be defined as FP/(FP+TN) x 100. The false positive (FP) results are from pregnancies with a SmartNIPT cfDNA test result positive for Down syndrome that are determined to be euploid after diagnostic testing or birth follow-up. True negatives (TN) will be defined as those pregnancies with a cfDNA test result negative for Down syndrome.
Down syndrome failure rate | Documentation of the failed result for Down syndrome will be considered confirmed when no results are returned for the second tested sample, typically within 14 days after enrollment.
  The cfDNA test failure rate will be computed using data from the general population (low) enrollment only (2,400 pregnancies) and be defined as TF/Total. The cfDNA initial test will be classified as an initial test failure (iTF), if the first sample tested fails to produce a complete set of interpretable results. All test failures will be followed by testing a second available sample, and if that is also unsuccessful in producing a complete set of interpretable results, it will be characterized as a test failure (TF).

SECONDARY OUTCOMES:
Trisomy 18 detection rate | Karyotype at chorionic villous sampling (CVS)/amniocentesis within 48 hours of enrollment OR at examination of products of conception if fetal loss up to 30 weeks post enrollment OR at newborn examination 24-48 hours after birth
  The cfDNA test detection rates for trisomy 18 will utilize both the general population (low risk) enrollment (2,400 pregnancies) as well as the high risk enrollment (250 pregnancies, all confirmed trisomy 21/18/13) and be defined as TP/(TP+FN). All low risk women with a cfDNA test positive for trisomy 18 will have comprehensive diagnostic follow-up as will all high risk women, assuring that all affected pregnancies in these two groups will have karyotype confirmation. The true positive (TP) SmartNIPT cfDNA test results will be positive and agree with the abnormal karyotype finding. The false negative (FN) SmartNIPT cfDNA test results will be negative for the abnormal karyotype finding.
Trisomy 13 detection rate | Karyotype at chorionic villous sampling (CVS)/amniocentesis within 48 hours of enrollment OR at examination of products of conception if fetal loss up to 30 weeks post enrollment OR at newborn examination 24-48 hours after birth
  The cfDNA test detection rates for trisomy 13 will utilize both the general population (low risk) enrollment (2,400 pregnancies) as well as the high risk enrollment (250 pregnancies, all confirmed trisomy 21/18/13) and be defined as TP/(TP+FN). All low risk women with a cfDNA test positive for trisomy 13 will have comprehensive diagnostic follow-up as will all high risk women, assuring that all affected pregnancies in these two groups will have karyotype confirmation. The true positive (TP) SmartNIPT cfDNA test results will be positive and agree with the abnormal karyotype finding. The false negative (FN) SmartNIPT cfDNA test results will be negative for the abnormal karyotype finding.
Trisomy 18 false positive rate | Karyotype at chorionic villous sampling (CVS)/amniocentesis within 48 hours of enrollment OR at examination of products of conception if fetal loss up to 30 weeks post enrollment. OR negative newborn examination 24-48 hours after birth
  The false positive rate for trisomy 18 will be computed using data from the general population (low risk) enrollment only (2,400 pregnancies) and be defined as FP/(FP+TN) x 100. The false positive (FP) results are from pregnancies with a SmartNIPT cfDNA test result positive for trisomy 18 that are determined to be euploid after diagnostic testing or birth follow-up. True negatives (TN) will be defined as those pregnancies with a cfDNA test result negative for trisomy 18.
Trisomy 13 false positive rate | Karyotype at chorionic villous sampling (CVS)/amniocentesis within 48 hours of enrollment OR at examination of products of conception if fetal loss up to 30 weeks post enrollment. OR negative newborn examination 24-48 hours after birth
  The false positive rate for trisomy 13 will be computed using data from the general population (low risk) enrollment only (2,400 pregnancies) and be defined as FP/(FP+TN) x 100. The false positive (FP) results are from pregnancies with a SmartNIPT cfDNA test result positive for trisomy 13 that are determined to be euploid after diagnostic testing or birth follow-up. True negatives (TN) will be defined as those pregnancies with a cfDNA test result negative for trisomy 13.
Trisomy 18 failure rate | Documentation of the failed result for Down syndrome will be considered confirmed when no results are returned for the second tested sample, typically within 14 days after enrollment.
  The cfDNA test failure rate will be computed using data from the general population (low) enrollment only (2,400 pregnancies) and be defined as TF/Total. The cfDNA initial test will be classified as an initial test failure (iTF), if the first sample tested fails to produce a complete set of interpretable results. All test failures will be followed by testing a second available sample, and if that is also unsuccessful in producing a complete set of interpretable results, it will be characterized as a test failure (TF).
Trisomy 13 failure rate | Documentation of the failed result for Down syndrome will be considered confirmed when no results are returned for the second tested sample, typically within 14 days after enrollment.
  The cfDNA test failure rate will be computed using data from the general population (low) enrollment only (2,400 pregnancies) and be defined as TF/Total. The cfDNA initial test will be classified as an initial test failure (iTF), if the first sample tested fails to produce a complete set of interpretable results. All test failures will be followed by testing a second available sample, and if that is also unsuccessful in producing a complete set of interpretable results, it will be characterized as a test failure (TF).
Fetal sex detection rate | Karyotype at chorionic villous sampling (CVS)/amniocentesis within 48 hours of enrollment OR at examination of products of conception if fetal loss up to 30 weeks post enrollment OR at newborn examination 24-48 hours after birth
  The cfDNA test detection rate for fetal sex will utilize only the general population (low risk) enrollment (2,400 pregnancies) and be defined as TP/(TP+FN) where the male sex is the target of testing (singleton pregnancies only). All low risk women will have the results of a clinical cfDNA test available to compare with the study's test. The fetal sex result on the clinical test will be considered the gold standard. True positive results will occur when the new test agrees with the clinical test result that the fetus is male. False negative results will occur when the clinical test reports male while the study's test reports female. In any instance where the two tests report discordant results for fetal sex, pregnancy follow-up (either via 2nd trimester ultrasound or birth examination) will resolve the discrepancy.
Fetal sex detection false positive rate | Karyotype at chorionic villous sampling (CVS)/amniocentesis within 48 hours of enrollment OR at examination of products of conception if fetal loss up to 30 weeks post enrollment. OR newborn examination 24-48 hours after birth reveal female sex
  The false positive rate for fetal sex will be computed using data from the general population (low risk) enrollment only (2,400 pregnancies) and be defined as FP/(FP+TN) x 100 where the male sex is the target of testing (singleton pregnancies only). All low risk women will have the results of a clinical cfDNA test available to compare with the study's test. The fetal sex result on the clinical test will be considered the gold standard. False positive (FP) results will occur when the study's cfDNA test predicts a male fetus in a pregnancy where female fetal sex is determined by clinical cfDNA testing. In any instance where the two tests report discordant results for fetal sex, pregnancy follow-up (either via 2nd trimester ultrasound or birth examination) will resolve the discrepancy. True negatives (TN) will be defined as those pregnancies where both clinical cfDNA test results and the study's DNA test results are negative for male sex.
Fetal sex detection failure rate | Documentation of the failed result for Down syndrome will be considered confirmed when no results are returned for the second tested sample, typically within 14 days after enrollment.
  The cfDNA test failure rate will be computed using data from the general population (low) enrollment only (2,400 pregnancies) and be defined as TF/Total. The cfDNA initial test will be classified as an initial test failure (iTF), if the first sample tested fails to produce a complete set of interpretable results. All test failures will be retested using a second sample and if that fails to produce a complete set of interpretable results, it will be counted as a test failure (TF).
Documentation of resources needed to implement SmartNIPT | Through study completion, 2 years.
  Determination of effort needed by non-molecular lab staff to implement SmartNIPT technology, costs and effort associated with bringing this non-NGS methodology into a non-molecular laboratory, and effort required to maintain proficiency in a clinical laboratory.

OTHER OUTCOMES:
Develop a post-hoc statistical algorithm suitable for expanded use of SmartNIPT | 2 months after confirmation of birth outcome of outstanding cases
  Based on the results of the VALUE Study, we intend to develop an algorithm that can be used to classify results and, if possible, assign reliable and validated patient-specific risks for Down syndrome, trisomy 18, trisomy 13, and prediction of fetal sex..

CONTACTS AND LOCATIONS:
Overall Officials: Glenn E Palomaki, PhD, Principal Investigator — Women and Infants Hospital of Rhode Island
Locations (16):
- United States (13):
  - Center for Fetal Medicine, Los Angeles, California
  - University of Colorado, Aurora, Colorado
  - Bridgeport Hospital, Bridgeport, Connecticut
  - University of South Florida, Tampa, Florida
  - Northwestern Memorial Medical Center, Chicago, Illinois
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - South Shore Hospital, South Weymouth, Massachusetts
  - Womens Health Care Group, Oaks, Pennsylvania
  - Magee Womens Hospital, Pittsburgh, Pennsylvania
  - Women & Infants Hospital of Rhode Island, Providence, Rhode Island
  - University of Texas, Houston, Texas
  - Swedish Medical Center, Seattle, Washington
- Canada (2):
  - North York General Hospital, Toronto, Ontario
  - GenoScience Diagnostic, Québec, Quebec
- University of Genoa - Hospital San Martino, Genova, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Dahl F, Ericsson O, Karlberg O, Karlsson F, Howell M, Persson F, Roos F, Stenberg J, Ahola T, Alftren I, Andersson B, Barkenas E, Brandner B, Dahlberg J, Elfman S, Eriksson M, Forsgren PO, Francois N, Gousseva A, Hakamali F, Janfalk-Carlsson A, Johansson H, Lundgren J, Mohsenchian A, Olausson L, Olofsson S, Qureshi A, Skarpas B, Savneby A, Astrom E, Ohman O, Westgren M, Kopp-Kallner H, Fianu-Jonasson A, Syngelaki A, Nicolaides K. Imaging single DNA molecules for high precision NIPT. Sci Rep. 2018 Mar 14;8(1):4549. doi: 10.1038/s41598-018-22606-0. PMID 29540801
- [Background] Ericsson O, Ahola T, Dahl F, Karlsson F, Persson F, Karlberg O, Roos F, Alftren I, Andersson B, Barkenas E, Boghos A, Brandner B, Dahlberg J, Forsgren PO, Francois N, Gousseva A, Hakamali F, Janfalk-Carlsson A, Johansson H, Lundgren J, Mohsenchian A, Olausson L, Olofsson S, Qureshi A, Skarpas B, Svahn P, Savneby A, Astrom E, Sahlberg A, Fianu-Jonasson A, Gautier J, Costa JM, Jacobsson B, Nicolaides K. Clinical validation of a novel automated cell-free DNA screening assay for trisomies 21, 13, and 18 in maternal plasma. Prenat Diagn. 2019 Oct;39(11):1011-1015. doi: 10.1002/pd.5528. Epub 2019 Aug 19. PMID 31429096
- [Result] Palomaki GE, Eklund EE, Kloza EM, Lambert-Messerlian GM. Assessment of a Simplified Cell-Free DNA Method for Prenatal Down Syndrome Screening. Clin Chem. 2022 Nov 3;68(11):1449-1458. doi: 10.1093/clinchem/hvac131. PMID 36103259